CLINICAL TRIAL: NCT07001501
Title: A Clinical Study of the Interactions Between Azvudine Tablets (FNC) and Itraconazole Capsules (ICZ)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KHYQZX-022-2021
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Azvudine
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 : FNC+ICZ;FNC;ICZ (Experimental)
  Interventions: Drug: Azvudine tablets(FNC) and Itraconazole Capsules (ICZ)
- Group 2 : ICZ;FNC+ICZ; FNC (Experimental)
  Interventions: Drug: Azvudine tablets(FNC) and Itraconazole Capsules (ICZ)
- Group 3 : FNC; ICZ; FNC+ICZ (Experimental)
  Interventions: Drug: Azvudine tablets(FNC) and Itraconazole Capsules (ICZ)

INTERVENTIONS:
Drug: Azvudine tablets(FNC) and Itraconazole Capsules (ICZ) — This study consisted of 3 cycles, each cycle was administered orally for 10 consecutive days, and the washout period between each cycle was 14 days. Subjects were administered the drug as follow:
  FNC 3 mg (1 tablet)+ICZ 200 mg (2 capsules) (taken at the same time), 1 time a day, orally, for 10 consecutive days; FNC: 3 mg (1 tablet) each time, 1 time a day, orally, for 10 consecutive days; ICZ: 200 mg (2 capsules) each time, 1 time a day, orally, for 10 consecutive days.
  Arms: Group 1 : FNC+ICZ;FNC;ICZ
Drug: Azvudine tablets(FNC) and Itraconazole Capsules (ICZ) — This study consisted of 3 cycles, each cycle was administered orally for 10 consecutive days, and the washout period between each cycle was 14 days. Subjects were administered the drug as follow:
  ICZ: 200 mg (2 capsules) each time, 1 time a day, orally, for 10 consecutive days; FNC 3 mg (1 tablet)+ICZ 200 mg (2 capsules) (taken at the same time), 1 time a day, orally, for 10 consecutive days; FNC: 3 mg (1 tablet) each time, 1 time a day, orally, for 10 consecutive days.
  Arms: Group 2 : ICZ;FNC+ICZ; FNC
Drug: Azvudine tablets(FNC) and Itraconazole Capsules (ICZ) — This study consisted of 3 cycles, each cycle was administered orally for 10 consecutive days, and the washout period between each cycle was 14 days. Subjects were administered the drug as follow:
  FNC: 3 mg (1 tablet) each time, 1 time a day, orally, for 10 consecutive days; ICZ: 200 mg (2 capsules) each time, 1 time a day, orally, for 10 consecutive days; FNC 3 mg (1 tablet)+ICZ 200 mg (2 capsules) (taken at the same time), 1 time a day, orally, for 10 consecutive days.
  Arms: Group 3 : FNC; ICZ; FNC+ICZ

SUMMARY:
Azvudine(FNC)，a nucleoside reverse transcriptase inhibitor, make itself a better candidate to be co-formulated in other anti-HIV therapies, thus to improve patient's compliance. FNC is a broad-spectrum RNA virus inhibitor that inhibits the novel coronavirus RNA-dependent RNA polymerase (RdRp).

This is a clinical study to evaluate the Interactions between Azvudine Tablets (FNC) and Itraconazole Capsules (ICZ) in healthy subjects. This is a single-center, randomized, open-label, three-cycles, three-treatment crossover clinical trial. Subjects was administered orally for 10 consecutive days each cycle, and the washout period between each cycle was 14 days. Biological sample collection and safety examination were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18 years or older (including 18 years) with an appropriate ratio of male to female participants;
2. The weight of men should be ≥ 50.0kg, and the weight of women should be ≥ 45.0kg. Body mass index (BMI) within the range of 19.0-26.0 (including the critical value).;
3. All fertile male and female subjects agreed to take appropriate and effective physical contraceptive measures from the screening period until the end of the trial, and to use effective physical and/or pharmacological contraceptive measures for 6 months after the trial ends, with no plans for sperm or egg donation;
4. Subjects fully understand the purpose, nature, process of the trial, and the potential adverse reactions, voluntarily agree to participate as subjects, and sign an informed consent form prior to the commencement of all study procedures;
5. Subjects must be able to communicate effectively with the researchers and understand and comply with all requirements of this study.

Exclusion Criteria:

1. Individuals with allergic constitutions, a history of drug or food allergies, especially those allergic to any components of this product and its excipients;
2. Individuals with a previous history of hypoglycemia;
3. Individuals who have abnormal results from physical examinations, vital signs check, clinical laboratory tests, 12-lead electrocardiograms, and other pre-trial relevant examinations, deemed clinically significant by the clinical researcher, and considered unqualified (normal reference range for vital signs: systolic blood pressure <90 mmHg or >140 mmHg, diastolic blood pressure <60 mmHg or >90 mmHg; pulse <60 bpm or >100 bpm);
4. Individuals with a history of alcohol abuse within the 12 months prior to screening (consuming ≥14 units of alcohol weekly: 1 unit = 285 ml of beer, or 25 ml of spirits, or 150 ml of wine) or those with positive alcohol breath test results before enrollment (test value >0 mg/100 ml);
5. Individuals with a history of drug abuse or use of illicit substances within the 12 months prior to screening, including repeated or excessive use of various anesthetics and psychoactive substances, addictive drugs [MDMA (Ecstasy), Methamphetamine (Ice), Ketamine, Morphine, THC (Marijuana)] or those with a positive result on the five-panel drug test before enrollment;
6. Individuals who had undergone surgery within 3 months prior to screening, especially those who had surgeries affecting drug absorption, distribution, metabolism, or excretion, or who plan to undergo surgery during the study;
7. Individuals who had used any drug that interacts with the trial medication within 30 days prior to screening, such as methadone, disopyramide, dofetilide, dronedarone, quinidine, ergot alkaloids (such as dihydroergotamine, ergometrine, ergotamine, methylergometrine), irinotecan, lurasidone, oral midazolam, pimozide, triazolam, felodipine, nisoldipine, ranolazine, eplerenone, cisapride, lovastatin, simvastatin, ticagrelor, CYP3A4 medium or strong inducers such as levoacemesadol, halofantrine, astemizole, imidolastine, terfenadine, serindole, benzylprodil, lecadipine, ivabradidine, domperidone and other CYP3A4 medium or strong inducers or CYP3A4/P-glycoprotein/BCRP substrates and erythromycin, azithromycin, levoxacin, etc.;
8. Individuals with a past medical history of cardiovascular, liver, kidney, pulmonary, gastrointestinal, neurological diseases, particularly any surgical conditions or diseases that might affect drug absorption, distribution, metabolism, and excretion, or conditions that could pose risks to trial participants;
9. Individuals with a history of mental illness (e.g., anxiety, depression);
10. Individuals with febrile illnesses within 3 days prior to screening;
11. Individuals who had received a novel coronavirus vaccine within 14 days prior to screening or received any other vaccine within 3 months prior to screening, or planed to receive a vaccine during the study;
12. Individuals who had participated in other clinical trials and received medication within 3 months prior to screening;
13. Individuals who consumed excessive amounts of tea, coffee, and/or beverages rich in caffeine, theobromine, and alcohol (more than 8 cups, with 1 cup = 250 ml) within 3 months prior to screening;
14. Individuals who had used any prescription medications, over-the-counter drugs, herbal medicines, dietary supplements, and functional vitamins within 14 days before the first dose;
15. Individuals who smoked an average of more than 5 cigarettes daily within 3 months prior to the first dose;
16. Individuals who had donated blood or experienced significant blood loss (greater than 400 ml, excluding normal physiological bleeding in women) within 3 months prior to the first dose, or who planed to donate blood or blood components during the study or within one week after the study;
17. Females who tested positive for pregnancy; pregnant or breastfeeding women; female participants who engaged in unprotected sexual intercourse with a partner within 14 days prior to the trial;
18. Individuals with poor conditions for vascular puncture, or who could not tolerate venous blood sampling, and/or had a history of vasovagal syncope;
19. Individuals deemed unsuitable for this study by the investigator.

(19) Individuals deemed unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Plasma Concentration at Steady State (Cmax, ss) of Azvudine and Itraconazole | Blood samples were collected on Day 8, 9, 10, 31, 32, 33, 54, 55 and 56 of the study.
Pharmacokinetics (PK): Time to Maximum Plasma Concentration at Steady State (Tmax, ss) of Azvudine and Itraconazole | Blood samples were collected on Day 8, 9, 10, 31, 32, 33, 54, 55 and 56 of the study.
Pharmacokinetics (PK): Elimination of Terminal Half-Life (t1/2) of Azvudine and Itraconazole | Blood samples were collected on Day 8, 9, 10, 31, 32, 33, 54, 55 and 56 of the study.

SECONDARY OUTCOMES:
Occurrence of Adverse Events | From enrollment to the end of the study on Day 59.
  Clinical presentation characteristics, severity, onset time, duration of adverse events, management measures, outcomes, and the correlation with the investigational drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Clinical Trial Research Center of Dongguan Kanghua Hospital, Guangdong, China